CLINICAL TRIAL: NCT03872817
Title: Development and Piloting of a Psychoeducational Intervention to Promote Mental Health Literacy in Adolescents in a School Context
Brief Title: Psychoeducational Intervention to Promote Adolescents' Mental Health Literacy in a School Context
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Enfermagem de Coimbra (Other)
Responsible Party: Principal Investigator, Tânia Manuel Moço Morgado, Psychiatric and Mental Health Nurse, Escola Superior de Enfermagem de Coimbra
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 71/2015
Record Dates: First submitted 2019-02-11; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Health Literacy
Keywords: Mental Health; Health Literacy; Adolescent; Schools
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants are assigned in two groups, an experimental group who will receive the psychoeducational intervention "ProLiSMentAl" and a control group who have usual intervention
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention ProLiSMentAl (Experimental): Experimental Group receive mental health literacy psychoeducational intervention called "ProLiSMentAl" that consist of 4 sessions of 90 minutes.
  Interventions: Other: Intervention ProLiSMentAl
- Control Group (No Intervention): Control Group receive usual approach.

INTERVENTIONS:
Other: Intervention ProLiSMentAl — Using different methods and pedagogical techniques, mental health literacy psychoeducational intervention called "ProLiSMentAl" consist of 4 sessions of 90 minutes: 1) improvement social anxiety recognition; 2) prevention strategies; 3) self-help strategies; 4) knowledge of first aid strategies and 5) knowledge of professionals and treatments available.
  Arms: Intervention ProLiSMentAl

SUMMARY:
Mental Health Literacy was defined as knowledge and beliefs about mental disorders that aid in its recognition, management or prevention. Portugal is the European country with the highest prevalence of mental illness in the population (22.9%) and anxiety disorders are the most common (16.5%). Approximately 20% of children and adolescents suffer from some mental disorder and about 8% of adolescents aged 13 to 18 years have some anxiety disorders. Portugal School Health Program 2015 evidences the promotion of health literacy and anxiety as areas of intervention in adolescence. The investigators intend to know the feasibility of a psychoeducational intervention to promote adolescents' mental health literacy (MHL) about anxiety in a school context.

DETAILED DESCRIPTION:
Mental Health Literacy (MHL) was defined as knowledge and beliefs about mental disorders that aid in its recognition, management or prevention and include several components: recognition of disorders to facilitate help-seeking; knowledge of professional help and treatments available; knowledge of effective self-help strategies; knowledge and skills to give first aid and support to others, and knowledge of how to prevent mental disorders. MHL is not simply knowledge of mental health problems, it is knowledge linked to action which can benefit one's own mental health or that of others. Portugal is the European country with the highest prevalence of mental illness in the population (22.9%) and anxiety disorders are the most common (16.5%). Approximately 20% of children and adolescents suffer from some mental disorder and about 8% of adolescents aged 13 to 18 years have some anxiety disorders. In a Portugal recent study, anxiety predominated in 66.3% (930) adolescents between the ages of 13 and 17 who used the urgency of a pediatric hospital from 2011 to 2014. Portugal School Health Program (2015) evidences the promotion of health literacy and anxiety as areas of intervention in adolescence.

The objectives of this study are: identify adolescents' MHL about anxiety in school setting; design an psychoeducational intervention to promote adolescents' MHL about anxiety in school setting; validate the content of that intervention and evaluate its feasibility.

Research Method(s): Medical Research Council's (MRC) framework and CReDECI Checklist were applied on the development and evaluation of complex interventions using quantitative, qualitative and mixed methods. Ethical considerations have taken place.

Implementation Strategies for Findings: Development of psychoeducational intervention to promote adolescents' MHL about anxiety in school setting supported by Health Promotion Model of Pender; Conceptual Model of Health Literacy and Integrative Model of Behavioral Prediction. Systematic reviews about adolescents' MHL and about MHL interventions showed reduced mental health literacy of adolescents and suggest some methods and pedagogical techniques. We designed a mental health literacy psychoeducational intervention about anxiety on adolescents in a school context called "ProLiSMentAl" using different methods and pedagogical techniques, consist of 4 sessions of 90 minutes: 1) Improvement social anxiety recognition; 2) prevention strategies; 3) self-help strategies; 4) knowledge of first aid strategies and 5) knowledge of professionals and treatments available. Contextual factors and determinants of the setting in the modelling of the intervention were given by a focus group with 6 health and education experts and a focus group with 6 adolescents and an e-delphi with 25 experts. After nurses' training and preparation meetings, mixed studies were carried out to model the final intervention and determine feasibility, acceptability and practicability of this complex intervention: 1) feasibility study: pre-experimental, before and after, without control group with 11 adolescents; 2) adolescents', health and education professionals' evaluation; 3) pilot study: quasi-experimental, before, after and 1month follow-up (n=21) with an equivalent control group (n=17).

ELIGIBILITY:
Inclusion Criteria:

All adolescents', students from 9th grade with informed consent.

Exclusion Criteria:

* students with special needs;
* students of other years of schooling
* students without informed consent.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2016-03-13 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of a psychoeducational intervention to promote adolescents' mental health literacy about anxiety in school setting using mental health literacy questionnaires. | Before, immediately following the psychoeducational intervention and 1 month follow-up
  Improvement and change of adolescents' mental health literacy from baseline, measured before, immediately following the psychoeducational intervention and 1 month follow-up.
  Measuring instruments: Mental Health Literacy Questionnaire.
  Treatment and analysis of data: content analysis and IBM SPSS Statistics 24.0

CONTACTS AND LOCATIONS:
Overall Officials: Tânia Morgado, RN, MSc, Principal Investigator — CHUC, EPE, EsenfC and UICISA:E

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jorm AF, Korten AE, Jacomb PA, Christensen H, Rodgers B, Pollitt P. "Mental health literacy": a survey of the public's ability to recognise mental disorders and their beliefs about the effectiveness of treatment. Med J Aust. 1997 Feb 17;166(4):182-6. doi: 10.5694/j.1326-5377.1997.tb140071.x. PMID 9066546
- [Background] Jorm AF. Improving the mental health of the population: where to next? Med J Aust. 2014 Jul 7;201(1):23-4. doi: 10.5694/mja14.00509. No abstract available. PMID 24999880
- [Background] Jorm AF. Mental health literacy: empowering the community to take action for better mental health. Am Psychol. 2012 Apr;67(3):231-43. doi: 10.1037/a0025957. Epub 2011 Oct 31. PMID 22040221
- [Background] Jorm AF. Mental health literacy. Public knowledge and beliefs about mental disorders. Br J Psychiatry. 2000 Nov;177:396-401. doi: 10.1192/bjp.177.5.396. PMID 11059991
- [Background] Loureiro LM. Questionnaire for Assessment of Mental Health Literacy - QuALiSMental: study of psychometric properties. Revista de Enfermagem Referência serIV(4): 79-88, 2015. https://dx.doi.org/10.12707/RIV14031
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M. Developing and evaluating complex interventions: the new Medical Research Council guidance. Int J Nurs Stud. 2013 May;50(5):587-92. doi: 10.1016/j.ijnurstu.2012.09.010. Epub 2012 Nov 15. No abstract available. PMID 23159157
- [Derived] Morgado T, Loureiro L, Rebelo Botelho MA, Marques MI, Martinez-Riera JR, Melo P. Adolescents' Empowerment for Mental Health Literacy in School: A Pilot Study on ProLiSMental Psychoeducational Intervention. Int J Environ Res Public Health. 2021 Jul 29;18(15):8022. doi: 10.3390/ijerph18158022. PMID 34360315